CLINICAL TRIAL: NCT04885595
Title: Bronchoscopic Diagnosis of Peripheral Lung Nodules Using Endobronchial Ultrasound Guided Forceps and Cryobiopsy. A Randomized-controlled Trial
Brief Title: Diagnosis of Peripheral Lung Nodules Using Cryobiopsy
Acronym: Cryo-Nodule
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Carolin Steinack, Principal Investigator, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2021-00323
Record Dates: First submitted 2021-04-18; First posted 2021-05-13 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Lung; Node
Keywords: Cryobiopsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forceps-Cryo 1.1 mm (Active Comparator): Forceps biopsy following cryobiopsy with a 1.1mm cryoprobe are obtained within the same session
  Interventions: Procedure: Forceps biopsy and cryobiopsy
- Forceps-Cryo 1.7 mm (Active Comparator): Forceps biopsy following cryobiopsy with a 1.7mm cryoprobe are obtained within the same session
  Interventions: Procedure: Forceps biopsy and cryobiopsy

INTERVENTIONS:
Procedure: Forceps biopsy and cryobiopsy — Once the nodule is visualized by radial EBUS, the position of the probe in relation to the lesion is noted. Routinely, forceps biopsy and cryobiopsy are used serially in each patient within the same session.

SUMMARY:
Since the traditional radial endobronchial ultrasound guided biopsy technique of solitary pulmonary nodules using the forceps has several shortcomings, the purpose of this study is to investigate a new biopsy technique using the transbronchial cryobrobe

DETAILED DESCRIPTION:
This is a prospective randomized trial to assess diagnostic accuracy and safety of cryobiopsy using two different outer diameters. Included patients are 1:1 randomized to receive forceps biopsy following cryobiopsy with a 1.1mm or 1.7mm cryoprobe.

ELIGIBILITY:
Inclusion Criteria:

* Solitary pulmonary nodule with indication of bronchoscopic diagnostic approach
* Age between 18 and 90 years
* Written informed consent after participant's information

Exclusion Criteria:

* Age < 18 and > 90 years
* Lacking ability to form an informed consent (including impaired judgement, communi-cation barriers)
* Contraindication against bronchoscopy (e.g. co-morbidities)
* INR > 2 or Thrombocytes < 50000
* Double antiplatelet drugs (e.g. ASS and Clopidogrel) within 7 days before biopsy
* Anticoagulation with NOAK within 48 hours before biopsy
* Moderate or severe pulmonary hypertension (mPAP > 30 mmHg, RV/RA >30 mmHg)
* Tumors suspicious of endobronchial growth

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | up to 1 month
  The diagnostic yield of the malign lesions that we were able to visualise with EBUS in percentage

SECONDARY OUTCOMES:
Size of harvested tissue in millimeter | up to 1 month
  The biopsies are assessed for total size in millimeter
Size of malign tissue in millimeter | up to 1 month
  The biopsies are assessed for size of malign tissue in milimeter
Occurrence of bleeding events | up to 1 month
  Occurrence of bleeding events
Size of artifact-free alvoelar space in percentage | up to 1 month
  Size of artifact-free alvoelar space in percentage
Radial endobronchial utrasound probe orientation (excentric, concentric, adjacent) | 1 day
  Lesion orientation with regards of the radial endobronchial ultrasound probe
Occurence of pneumothorax | up to 1 month
  Detection with X-ray

CONTACTS AND LOCATIONS:
Overall Officials: Carolin Steinack, MD, Principal Investigator — University of Zurich
Locations (1):
- University hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No